CLINICAL TRIAL: NCT07094711
Title: Safety, Immunogenicity, and Efficacy of Therapeutic Mycobacterium Bovis BCG in Patients With Mycobacterium Avium Complex Lung Disease (BOOST)
Brief Title: Safety, Immunogenicity, and Efficacy of Therapeutic Mycobacterium Bovis BCG (BOOST)
Acronym: BOOST
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Eric R. Houpt, MD, Professor and Chief, Division of Infectious Diseases and International Health, Medicine: Infectious Diseases and International Health, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 302296Boost
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Mycobacterium Avium-intracellulare Infection; Mycobacterium Infections, Nontuberculous
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; Mycobacterium Infections, Nontuberculous | interventions — Vaccines; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Standard two-sample comparisons will be used to compare changes in immunogenicity.
  The number and type of adverse events will be tabulated by treatment group. Chi-squared tests will be used to compare the groups on the proportion of patients in each group experiencing severe adverse events. Standard one-side, two-sample confidence intervals will be used to summarize the difference in proportions between the groups.
  Logistic regression with generalized estimating equations (GEE) will be used for the proportion of monthly sputum cultures positive for MAC after BCG vaccination or placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active BCG (Active Comparator): Biological/Vaccine: Mycobacterium bovis Bacillus Calmette Guerin (BCG) vaccine
  Interventions: Biological: Mycobacterium bovis Bacillus Calmette Guerin (BCG) vaccine
- Placebo (Placebo Comparator): preservative-free saline
  Interventions: Drug: preservative-free saline

INTERVENTIONS:
Biological: Mycobacterium bovis Bacillus Calmette Guerin (BCG) vaccine — Subjects will be randomized to a single intradermal injection of BCG or placebo vaccine.
  Participants randomized to the BCG arm will receive TICE® BCG. Freeze-dried vaccine is produced in vials, each containing 1 to 8 x^108 colony forming units (CFU). A vial will be reconstituted in 20 mL of preservative-free saline. Administration of 0.1 mL will contain ~2x^106 CFU, which accounts for approximately 0.25 mg of the attenuated Mycobacterium bovis. Administration of 0.1 mL of diluted vaccine will be given per dose, intradermally.
  Other Names: TICE® BCG
  Arms: Active BCG
Drug: preservative-free saline — Patients randomized to the placebo arm will receive 0.1 mL preservative-free saline alone.
  Other Names: saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out if the Mycobacterium bovis Bacillus Calmette Guerin (BCG) vaccine can be used safely to treat Mycobacterium avium complex (MAC) lung disease.

Researchers will compare responses from patients with MAC lung disease after receiving an injection of BCG or placebo (a look-alike substance that contains no drug)

Participants in the study:

* Receive a BCG or placebo injection at UVA study center on Day 0
* Come to UVA study center on Day 60
* Come to UVA study center at the end of the study
* Answer surveys and questionnaires about how you are doing
* Have blood drawn 3 times, on injection day, day 60, and at end of study
* Give the study team personal and demographic information
* Discuss any new symptoms with the study team
* Provide monthly sputum samples per usual care

DETAILED DESCRIPTION:
Mycobacterium avium complex (MAC) lung disease (LD) is an increasingly prevalent condition in the United States. Treatment involves administration of multiple antibiotics for at least 12 months and many patients still fail, or infection recurs. New therapeutic strategies are needed. We hypothesize that Mycobacterium bovis Bacillus Calmette Guerin (BCG) will have microbiologic activity against MAC during lung disease, because of

* Its mycobacterium antigens shared with MAC (1).
* In vitro evidence that BCG stimulates MAC-specific immune responses in mice and humans (2, 3).
* In vivo evidence that BCG reduces MAC in mice with established infection (4). Clinical evidence for BCG protection against MAC infection in HIV patients and in children (5, 6).

Objectives:

The primary objective is to determine the safety and immunogenicity of BCG against MAC lung disease after intradermal vaccination with BCG or placebo.

The secondary objectives include:

* the microbiologic efficacy of BCG compared to placebo.
* to determine if BCG is superior to placebo in reducing all-cause respiratory illness requiring additional antibiotics, healthcare assessment, or admission.

Endpoints:

Primary endpoints:

* Safety and tolerability of intradermal BCG (TICE®) in this patient population, compared to placebo, assessed by weekly questionnaire of adverse events over 12 weeks.
* Serious adverse events related to the intradermal BCG over 12 months.
* Immunogenicity of BCG as measured by the change in BCG-induced IFN-γ production in PBMCs 60 days after vaccination, compared to placebo.

Secondary endpoints:

* Proportion of monthly sputum cultures positive for MAC after BCG vaccine or placebo over 24 months.
* Immunogenicity of BCG on MAC-specific IFN-γ responses.
* Proportion of patients with MAC culture conversion and MAC recurrence within 24 months.
* Rates of all-cause respiratory illness requiring additional antibiotics, healthcare assessment, or admission over 24 months.
* Symptom scores using the Quality of Life- Bronchiectasis Respiratory (QOL-BR) questionnaire over 24 months.
* Adverse Events of Special Interest (local/systemic M. bovis BCG infection) over 24 months.

Exploratory endpoints:

* Assess the efficacy of BCG versus placebo on chest imaging score.
* While the study is not powered to detect differences among subgroups, we will enumerate whether above endpoints are modified among these patient subgroups: cavitary versus non-cavitary disease, age, gender, the species of MAC infection, and those with higher IFN-γ responses.
* Assess PBMC cytokine responses beyond IFN-γ.
* Assess durability of immune responses at 24 months.

Study Population:

We aim to enroll a total of 48 participants with MAC, of which 24 will be randomized to receive each of BCG and placebo.

ELIGIBILITY:
Inclusion Criteria

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Male or female aged ≥18 years
2. Mycobacterium avium complex lung disease as evidenced by diagnosis or treatment for MAC lung disease by pulmonologist or infectious disease physician in the medical record. The following data will be extracted from the medical record:

   1. History of at least 2 MAC positive respiratory cultures, one of which is within 1 year of enrollment. In the event a MAC positive culture is from bronchial lavage or biopsy, one culture rather than 2 will meet criteria.
   2. Respiratory and/or constitutional symptoms consistent with MAC lung disease
   3. Nodular or cavitary opacities on chest radiograph or bronchiectasis with multiple small nodules on high-resolution computed tomography
3. Provision of signed and dated informed consent form
4. Stated willingness to comply with all study procedures
5. Women of childbearing potential (WOCBP) (i.e., fertile following menarche and until becoming postmenopausal unless permanently sterile) agree to practice a highly effective method of birth control from Day 0 to at least 90 days after study intervention. Some examples of acceptable birth controls are:

   1. True abstinence (refraining from heterosexual intercourse during the entire study),
   2. Copper intrauterine device (IUD),
   3. Hormonal methods (levonorgestrel-releasing intrauterine system, progestogen implant, combined oral contraceptive pill [combined with barrier method]), exclusive homosexual relationship) sole male partner who has undergone surgical sterilization

Exclusion Criteria

Selection of study participants will be equitable, but an individual who meets any of the following criteria will be excluded from participation in this study:

1. Currently receiving antibiotics prescribed for their MAC lung disease
2. Having received any antibacterial antibiotics within the past 14 days prior to study vaccination, day 0
3. Known allergy, intolerance or other contraindication to isoniazid or rifampin or ethambutol
4. Expectation of starting anti-MAC lung disease antibiotics in the next 2 months per patient or their physician
5. Persons with congenital or acquired immune deficiencies (e.g., HIV infection; leukemia, lymphoma, or cancer therapy within the past 2 years; immunosuppressive therapy such as anti B cell depleting therapies, corticosteroids (>20 mg/day for > 14 days), dupilumab, elivaldogene, etrasimod, cytotoxic chemotherapy, miscellaneous oncologic agents, therapeutic immunosuppressant agents, methotrexate, teplizumab, tezepelumab, tildrakizumab, tralokinumab, ustekinumab). Persons with lung and other solid organ transplants/hematologic stem cell transplants who may be contraindicated to receive a live vaccine. Point of care HIV testing must be negative at baseline.
6. Prior BCG Vaccination. If unknown Bcgatlas.org shall be consulted for local vaccination administration policies.
7. Known pregnancy at the time of screening or breastfeeding at the time of enrollment (pregnancy test negative at baseline if applicable)
8. Cystic fibrosis
9. Active tuberculosis: Active tuberculosis (respiratory AFB culture growing Mycobacterium tuberculosis complex within the past 4 months).
10. Known exposure to a case of active pulmonary tuberculosis within 10 weeks of enrollment
11. Known prior hypersensitivity reaction to BCG or any component of the BCG vaccine
12. Received live injectable vaccine within 28 days of day 0 study vaccination
13. Any condition in the opinion of the investigator that may confound the study endpoints Note that colonization or co-infection with other nontuberculous mycobacteria is not exclusionary, as MAC will be the endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 12 weeks after intervention
  Safety and tolerability of intradermal BCG (TICE®) in this patient population, compared to placebo, assessed by weekly questionnaire of adverse events. Licensed study team member will follow-up on any events reported to be more than mild. Follow-up will be completed as a telemedicine or in person visit
Serious adverse events | 12 months
  Serious adverse events related to the intradermal BCG over 12 months after intervention.
Immunogenicity | 24 months
  Compare changes in immunogenicity, as measured by IFN-gamma production between the BCG and placebo groups. We will assess for increases in T cell immune responses against BCG and MAC, as measured by cytokine production, in those who received the BCG vaccine and those that received placebo. We will use ex vivo T cell stimulation assays to quantify the antigen specific T cell responses and assess cytokine production via flow cytometry and/or multiplexed enzyme-linked immunosorbent assay (Luminex).

SECONDARY OUTCOMES:
Sputum cultures | 24 months
  Compare proportion of sputum cultures positive for MAC between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia Health, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Every attempt will be made to publish results in peer-reviewed journals. Data from this study may be requested from other researchers 2 years after the publication date of the primary endpoint by contacting Dr. Houpt. No protected health information will be shared.

REFERENCES:
- [Background] Blazevic A, Edwards RL, Xia M, Eickhoff CS, Hamzabegovic F, Meza KA, Ning H, Tennant J, Mosby KJ, Ritchie JC, Girmay T, Lai L, McCullough M, Beck A, Kelley C, Edupuganti S, Kabbani S, Buchanan W, Makhene MK, Voronca D, Cherikh S, Goll JB, Rouphael NG, Mulligan MJ, Hoft DF. Phase 1 Open-Label Dose Escalation Trial for the Development of a Human Bacillus Calmette-Guerin Challenge Model for Assessment of Tuberculosis Immunity In Vivo. J Infect Dis. 2024 May 15;229(5):1498-1508. doi: 10.1093/infdis/jiad441. PMID 38019956
- [Background] Allen HF, Klingensmith GJ, Jensen P, Simoes E, Hayward A, Chase HP. Effect of Bacillus Calmette-Guerin vaccination on new-onset type 1 diabetes. A randomized clinical study. Diabetes Care. 1999 Oct;22(10):1703-7. doi: 10.2337/diacare.22.10.1703. PMID 10526739
- [Background] Bricks LF. [Percutaneous or intradermal BCG vaccine?]. J Pediatr (Rio J). 2004 Mar-Apr;80(2):93-8. Portuguese. PMID 15079177
- [Background] Roy A, Eisenhut M, Harris RJ, Rodrigues LC, Sridhar S, Habermann S, Snell L, Mangtani P, Adetifa I, Lalvani A, Abubakar I. Effect of BCG vaccination against Mycobacterium tuberculosis infection in children: systematic review and meta-analysis. BMJ. 2014 Aug 5;349:g4643. doi: 10.1136/bmj.g4643. PMID 25097193
- [Background] Koekenbier EL, Fohse K, van de Maat JS, Oosterheert JJ, van Nieuwkoop C, Hoogerwerf JJ, Grobusch MP, van den Bosch MAAJ, van de Wijgert JHH, Netea MG, Rosendaal FR, Bonten MJM, Werkhoven CHHV; BCG-PRIME study group. Bacillus Calmette-Guerin vaccine for prevention of COVID-19 and other respiratory tract infections in older adults with comorbidities: a randomized controlled trial. Clin Microbiol Infect. 2023 Jun;29(6):781-788. doi: 10.1016/j.cmi.2023.01.019. Epub 2023 Feb 2. PMID 36736662
- [Background] Pittet LF, Messina NL, Orsini F, Moore CL, Abruzzo V, Barry S, Bonnici R, Bonten M, Campbell J, Croda J, Dalcolmo M, Gardiner K, Gell G, Germano S, Gomes-Silva A, Goodall C, Gwee A, Jamieson T, Jardim B, Kollmann TR, Lacerda MVG, Lee KJ, Lucas M, Lynn DJ, Manning L, Marshall HS, McDonald E, Munns CF, Nicholson S, O'Connell A, de Oliveira RD, Perlen S, Perrett KP, Prat-Aymerich C, Richmond PC, Rodriguez-Bano J, Dos Santos G, da Silva PV, Teo JW, Villanueva P, Warris A, Wood NJ, Davidson A, Curtis N; BRACE Trial Consortium Group. Randomized Trial of BCG Vaccine to Protect against Covid-19 in Health Care Workers. N Engl J Med. 2023 Apr 27;388(17):1582-1596. doi: 10.1056/NEJMoa2212616. PMID 37099341
- [Background] Dionato FAV, Jalalizadeh M, Buosi K, Visacri MB, Dal Col LSB, Giacomelli CF, Leme PAF, Maia CL, Moriel P, Reis LO. BCG vaccine safety in COVID-19 convalescent adults: BATTLE a randomized controlled trial. Vaccine. 2022 Jul 30;40(32):4603-4608. doi: 10.1016/j.vaccine.2022.06.039. Epub 2022 Jun 20. PMID 35738969
- [Background] Tsilika M, Taks E, Dolianitis K, Kotsaki A, Leventogiannis K, Damoulari C, Kostoula M, Paneta M, Adamis G, Papanikolaou I, Stamatelopoulos K, Bolanou A, Katsaros K, Delavinia C, Perdios I, Pandi A, Tsiakos K, Proios N, Kalogianni E, Delis I, Skliros E, Akinosoglou K, Perdikouli A, Poulakou G, Milionis H, Athanassopoulou E, Kalpaki E, Efstratiou L, Perraki V, Papadopoulos A, Netea MG, Giamarellos-Bourboulis EJ. ACTIVATE-2: A Double-Blind Randomized Trial of BCG Vaccination Against COVID-19 in Individuals at Risk. Front Immunol. 2022 Jul 5;13:873067. doi: 10.3389/fimmu.2022.873067. eCollection 2022. PMID 35865520
- [Background] Giamarellos-Bourboulis EJ, Tsilika M, Moorlag S, Antonakos N, Kotsaki A, Dominguez-Andres J, Kyriazopoulou E, Gkavogianni T, Adami ME, Damoraki G, Koufargyris P, Karageorgos A, Bolanou A, Koenen H, van Crevel R, Droggiti DI, Renieris G, Papadopoulos A, Netea MG. Activate: Randomized Clinical Trial of BCG Vaccination against Infection in the Elderly. Cell. 2020 Oct 15;183(2):315-323.e9. doi: 10.1016/j.cell.2020.08.051. Epub 2020 Sep 1. PMID 32941801
- [Background] Villanueva P, Crawford NW, Garcia Croda M, Collopy S, Araujo Jardim B, de Almeida Pinto Jardim T, Marshall H, Prat-Aymerich C, Sawka A, Sharma K, Troeman D, Wadia U, Warris A, Wood N, Messina NL, Curtis N, Pittet LF. Safety of BCG vaccination and revaccination in healthcare workers. Hum Vaccin Immunother. 2023 Aug 1;19(2):2239088. doi: 10.1080/21645515.2023.2239088. PMID 37551885
- [Background] Fritschi N, Curtis N, Ritz N. Bacille Calmette Guerin (BCG) and new TB vaccines: Specific, cross-mycobacterial and off-target effects. Paediatr Respir Rev. 2020 Nov;36:57-64. doi: 10.1016/j.prrv.2020.08.004. Epub 2020 Aug 20. PMID 32958428
- [Background] Zwerling A, Behr MA, Verma A, Brewer TF, Menzies D, Pai M. The BCG World Atlas: a database of global BCG vaccination policies and practices. PLoS Med. 2011 Mar;8(3):e1001012. doi: 10.1371/journal.pmed.1001012. Epub 2011 Mar 22. PMID 21445325
- [Background] Dow CT, Kidess L. BCG Vaccine-The Road Not Taken. Microorganisms. 2022 Sep 27;10(10):1919. doi: 10.3390/microorganisms10101919. PMID 36296196
- [Background] Greinert U, Schlaak M, Rusch-Gerdes S, Flad HD, Ernst M. Low in vitro production of interferon-gamma and tumor necrosis factor-alpha in HIV-seronegative patients with pulmonary disease caused by nontuberculous mycobacteria. J Clin Immunol. 2000 Nov;20(6):445-52. doi: 10.1023/a:1026407815946. PMID 11202234
- [Background] Gramegna A, Lombardi A, Lore NI, Amati F, Barone I, Azzara C, Cirillo D, Aliberti S, Gori A, Blasi F. Innate and Adaptive Lymphocytes in Non-Tuberculous Mycobacteria Lung Disease: A Review. Front Immunol. 2022 Jun 28;13:927049. doi: 10.3389/fimmu.2022.927049. eCollection 2022. PMID 35837393
- [Background] Winthrop K, Rivera A, Engelmann F, Rose S, Lewis A, Ku J, Bermudez L, Messaoudi I. A Rhesus Macaque Model of Pulmonary Nontuberculous Mycobacterial Disease. Am J Respir Cell Mol Biol. 2016 Feb;54(2):170-6. doi: 10.1165/rcmb.2015-0256RC. PMID 26562499
- [Background] Andersen P, Doherty TM. The success and failure of BCG - implications for a novel tuberculosis vaccine. Nat Rev Microbiol. 2005 Aug;3(8):656-62. doi: 10.1038/nrmicro1211. PMID 16012514
- [Background] Griffith DE, Eagle G, Thomson R, Aksamit TR, Hasegawa N, Morimoto K, Addrizzo-Harris DJ, O'Donnell AE, Marras TK, Flume PA, Loebinger MR, Morgan L, Codecasa LR, Hill AT, Ruoss SJ, Yim JJ, Ringshausen FC, Field SK, Philley JV, Wallace RJ Jr, van Ingen J, Coulter C, Nezamis J, Winthrop KL; CONVERT Study Group. Amikacin Liposome Inhalation Suspension for Treatment-Refractory Lung Disease Caused by Mycobacterium avium Complex (CONVERT). A Prospective, Open-Label, Randomized Study. Am J Respir Crit Care Med. 2018 Dec 15;198(12):1559-1569. doi: 10.1164/rccm.201807-1318OC. PMID 30216086
- [Background] Field SK, Fisher D, Cowie RL. Mycobacterium avium complex pulmonary disease in patients without HIV infection. Chest. 2004 Aug;126(2):566-81. doi: 10.1378/chest.126.2.566. PMID 15302746
- [Background] Adjemian J, Olivier KN, Seitz AE, Holland SM, Prevots DR. Prevalence of nontuberculous mycobacterial lung disease in U.S. Medicare beneficiaries. Am J Respir Crit Care Med. 2012 Apr 15;185(8):881-6. doi: 10.1164/rccm.201111-2016OC. Epub 2012 Feb 3. PMID 22312016
- [Background] Schildknecht KR, Pratt RH, Feng PI, Price SF, Self JL. Tuberculosis - United States, 2022. MMWR Morb Mortal Wkly Rep. 2023 Mar 24;72(12):297-303. doi: 10.15585/mmwr.mm7212a1. PMID 36952282
- [Background] Winthrop KL, Marras TK, Adjemian J, Zhang H, Wang P, Zhang Q. Incidence and Prevalence of Nontuberculous Mycobacterial Lung Disease in a Large U.S. Managed Care Health Plan, 2008-2015. Ann Am Thorac Soc. 2020 Feb;17(2):178-185. doi: 10.1513/AnnalsATS.201804-236OC. PMID 31830805
- [Background] Strollo SE, Adjemian J, Adjemian MK, Prevots DR. The Burden of Pulmonary Nontuberculous Mycobacterial Disease in the United States. Ann Am Thorac Soc. 2015 Oct;12(10):1458-64. doi: 10.1513/AnnalsATS.201503-173OC. PMID 26214350
- [Background] Orujyan D, Narinyan W, Rangarajan S, Rangchaikul P, Prasad C, Saviola B, Venketaraman V. Protective Efficacy of BCG Vaccine against Mycobacterium leprae and Non-Tuberculous Mycobacterial Infections. Vaccines (Basel). 2022 Mar 3;10(3):390. doi: 10.3390/vaccines10030390. PMID 35335022
- [Background] Zimmermann P, Finn A, Curtis N. Does BCG Vaccination Protect Against Nontuberculous Mycobacterial Infection? A Systematic Review and Meta-Analysis. J Infect Dis. 2018 Jul 24;218(5):679-687. doi: 10.1093/infdis/jiy207. PMID 29635431
- [Background] Rais M, Abdelaal H, Reese VA, Ferede D, Larsen SE, Pecor T, Erasmus JH, Archer J, Khandhar AP, Cooper SK, Podell BK, Reed SG, Coler RN, Baldwin SL. Immunogenicity and protection against Mycobacterium avium with a heterologous RNA prime and protein boost vaccine regimen. Tuberculosis (Edinb). 2023 Jan;138:102302. doi: 10.1016/j.tube.2022.102302. Epub 2022 Dec 27. PMID 36586154
- [Background] Abate G, Hamzabegovic F, Eickhoff CS, Hoft DF. BCG Vaccination Induces M. avium and M. abscessus Cross-Protective Immunity. Front Immunol. 2019 Feb 19;10:234. doi: 10.3389/fimmu.2019.00234. eCollection 2019. PMID 30837992
- [Background] Larsen SE, Reese VA, Pecor T, Berube BJ, Cooper SK, Brewer G, Ordway D, Henao-Tamayo M, Podell BK, Baldwin SL, Coler RN. Subunit vaccine protects against a clinical isolate of Mycobacterium avium in wild type and immunocompromised mouse models. Sci Rep. 2021 Apr 27;11(1):9040. doi: 10.1038/s41598-021-88291-8. PMID 33907221
- [Background] Harboe M, Mshana RN, Closs O, Kronvall G, Axelsen NH. Cross-reactions between mycobacteria. II. Crossed immunoelectrophoretic analysis of soluble antigens of BCG and comparison with other mycobacteria. Scand J Immunol. 1979;9(2):115-24. doi: 10.1111/j.1365-3083.1979.tb02713.x. PMID 106465